CLINICAL TRIAL: NCT00072150
Title: Phase II Trial of PS-341 (Bortezomib) in Patients With Previously Treated Advanced Urothelial Tract Transitional Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02787; CALGB-90207; U10CA031946 (NIH)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Bladder Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Stage III Bladder Cancer; Stage III Urethral Cancer; Stage IV Bladder Cancer; Stage IV Urethral Cancer; Transitional Cell Carcinoma of the Bladder; Ureter Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms; Ureteral Neoplasms | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Patients with a solitary site of disease (i.e., lung or nodal metastases) and who have a partial response (PR) may be considered for surgical resection. Patients with a PR with residual disease after salvage surgery are eligible to continue study therapy. Patients who achieve a complete response, either through resection or bortezomib therapy, receive 2 additional courses of study therapy.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. This phase II trial is studying how well bortezomib works in treating patients with advanced transitional cell carcinoma of the urothelium.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of PS-341 in patients with measurable advanced urothelial transitional cell carcinoma who have not responded to, or have relapsed after one prior conventional chemotherapy.

II. To determine the safety and toxicity of PS-341 administered in this group of patients.

III. To estimate duration of objective response, progression-free survival and overall survival in this group of patients.

OUTLINE: This is a multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with a solitary site of disease (i.e., lung or nodal metastases) and who have a partial response (PR) may be considered for surgical resection. Patients with a PR with residual disease after salvage surgery are eligible to continue study therapy. Patients who achieve a complete response, either through resection or bortezomib therapy, receive 2 additional courses of study therapy.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 15-40 patients will be accrued for this study within 13-17 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of transitional cell carcinoma (TCC) of the bladder, urethra, ureter or renal pelvis; histologic documentation of metastatic/recurrent disease is not required; clinical staging, but not pathological staging, is required
* All patients must have received only one prior systemic chemotherapy regimen for advanced or metastatic disease (which must have included at least one of the following chemotherapy agents: cisplatin, carboplatin, paclitaxel, docetaxel or gemcitabine), with progression documented during or after that treatment; neoadjuvant as well as adjuvant combination chemotherapy is considered a systemic chemotherapy; radiosensitizing single agent chemotherapy is not considered prior systemic therapy
* Patients must have completed radiotherapy (RT) or chemotherapy >= 4 weeks prior to registration on this trial; patients must have recovered from previous treatments or returned to their baseline in the judgment of the enrolling physician
* No Prior treatment with PS-341 or other proteasome inhibitors
* No prior treatment with investigational agents as single agent therapy; however, the incorporation of an investigational agent into the prior systemic chemotherapy regimen is allowed
* Patients must have measurable disease;

  * Measurable Disease is defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as >10 mm with spiral CT scan
  * Non-measurable disease: Patients with ONLY non-measurable disease are not eligible for this trial

    * Nonmeasurable disease is defined as all other lesions, including small lesions (longest diameter <20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions, which include the following:

      * Bone lesions;
      * Leptomeningeal disease;
      * Ascites;
      * Pleural/pericardial effusion;
      * Inflammatory breast disease;
      * Lymphangitis cutis/pulmonis;
      * Abdominal masses that are not confirmed and followed by imaging techniques;
      * Cystic lesions
      * Primary bladder masses
* CTC (ECOG) performance status =< 2
* Patients must have =< grade 1 peripheral neuropathy at baseline
* No known active brain metastases; patients may not have evidence of active brain metastases; screening CT or MRI is not required, unless there is clinical suspicion of brain metastases
* Pregnant and/or nursing women are not eligible for this trial as chemotherapy is thought to present substantial risk to the fetus/infant; men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while in this study; pregnant and/or nursing women are not eligible for this trial as chemotherapy is thought to present substantial risk to the fetus/infant; men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while in this study
* Creatinine =< 2.5 mg/dl or measured or calculated creatinine clearance > 30 ml/min)
* ALT and AST =< 2.5 x ULN
* Total bilirubin =< 1.8 mg/dL
* Granulocytes >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 8 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-10; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Response rates (CR+PR) determined according to the RECIST criteria | Up to 6 years
  95% confidence intervals will be computed using the binomial distribution.

SECONDARY OUTCOMES:
Duration of objective response | From the date of the first CR or PR to the date that the patient had disease progression (or death), assessed up to 6 years
  The Kaplan-Meier product-limit method will be used to estimate.
Toxicity by type, frequency, and severity | Up to 6 years
  95% confidence intervals for the toxicity rates will be computed using the binomial distribution.
Progression free survival | From the date of initiation of treatment to date of progression or death due to any cause, whichever occurs first, assessed up to 6 years
  The Kaplan-Meier product-limit method will be used to estimate.
Overall survival | From the date of initiation of treatment to date of death due to any cause, assessed up to 6 years
  The Kaplan-Meier product-limit method will be used to estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rosenberg, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- UCSF-Mount Zion, San Francisco, California, United States